CLINICAL TRIAL: NCT02130089
Title: Can Dietitians Reduce Interdialytic Weight Gain in at Risk Hemodialysis Patients Through Tailored Education on Dietary Sodium and Fluid Intake?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Alison Steiber, Chief Science Officer, Academy of Nutrition and Dietetics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-186
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: End Stage Renal Disease Requiring Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): Intensive tailored education
  Interventions: Behavioral: Intensive Tailored Education

INTERVENTIONS:
Behavioral: Intensive Tailored Education

SUMMARY:
The purpose of this project is to understand if more frequent education of dialysis patients (patients with kidney failure who get their blood cleaned and fluid removed by a machine instead of their kidneys) on reducing sodium intake reduces the amount of fluid weight that patients gain between dialysis sessions. Patients who usually gain more fluid than is considered ideal will be recruited for this project. Because all patients gain different amounts to start, data will be collected for 3 months while the patients receive their usual amount of dietitian education. Then the patients will receive intensive (2x/month) education on reducing sodium intake from the dietitian and the same data will be collected to see if they gain less after the education. After 3 months of intensive education, data will be collected for one more month to see if patients keep gaining less or if they go back to their old patterns.

ELIGIBILITY:
Inclusion Criteria:

* Average Interdialytic weight gain (IDWG) for 2 weeks prior to screening period greater than or equal to 4% estimated dry weight
* Able to sign the locally approved informed consent
* Willing to receive dietitian education on sodium and fluid control during normal dialysis time
* Receiving thrice weekly maintenance hemodialysis for greater than or equal to 6 months Age greater than or equal to 18 years

Exclusion Criteria:

* On hospice or international equivalent
* Receiving corticosteroid treatment
* Less than 18 years old
* On interdialytic parenteral nutrition
* Transfer to another facility expected within 3 months
* Severe malnutrition, as assessed by Subjective Global Assessment (SGA) or other standard assessment tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Average Percent Interdialytic Weight Gain | monthly for 7 months

SECONDARY OUTCOMES:
Thirst Intensity | monthly for 7 months
  will be measured by a 100 mm Visual Analog Scale. Patients are asked to mark the point on the VAS which represents their work thirst since the last dialysis. Zero is considered no thirst and 100 is extremely thirsty. This tool has been shown to correlate to the Thirst Distress tool developed by Welsh in 2002.
Sodium and Fluid Knowledge | Monthly for 4 months
  Will be assessed using the sodium questions of the tool created by Kim (Korean J Nutr 2001), as modified by Park (J Ren Nutr 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra McLellan, Principal Investigator — Auckland Board of Health
Locations (1):
- Auckland Board of Health, Auckland, New Zealand